CLINICAL TRIAL: NCT04755335
Title: Ultrasonic Perfusion Imaging of Peripheral Vascular Disease
Brief Title: Ultrasonic Perfusion Estimation in Calf Muscle
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Azra Alizad, Principal Investigator, Mayo Clinic
Other Study IDs: 19-002559; R01HL148664 (NIH); 5R01HL148664-02 (NIH)
Record Dates: First submitted 2021-02-02; First posted 2021-02-16 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Arterial Disease
Keywords: Blood flow; Blood Vessel; Ischemia; Calf muscle pain; Vascular; Ultrasound; Intermitant claudication; Cramp
MeSH Terms: conditions — Peripheral Arterial Disease; Ischemia; Muscle Cramp | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Early detection of PAD, assessment of the disease progression and treatment response: The objective of this arm of the study is to evaluate the potentials of Ultrasound Perfusion imaging technique for early detection of peripheral arterial disease in patients and assess the disease progression and monitor the treatment response.
  The investigators anticipate that our new cost-effective and non-invasive ultrasound perfusion technique offers a quantitative perfusion estimation of calf muscle that would separate PAD from non-PAD and help early detection of PAD and would help monitoring the disease progression and treatment response.
  Interventions: Diagnostic Test: Ultrasound
- Healthy volunteers: A group of healthy volunteers ages 18 and above with no history of smoking, cardiovascular, diabetes or surgery on legs.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — In this project, The investigators will use Alpinion ECUBE-12R (Alpinion, Bothell, WA) US platform. This state-of-the-art research US machine provides beam formed as well as Plane-Wave imaging options that allow high frame rate imaging. The investigators have characterized the acoustic output of this system for safe human studies and obtained the IRB approval for human studies. It should be noted that our technique is not limited to the Alpinion system; the investigators can also use other US systems, such as Verasonics, Vantage, (Redmond, WA). This technique can be adapted to other modern US machines in the future.

SUMMARY:
The purpose of this study is to evaluate the potential of ultrasound perfusion imaging technique for assessing the progression of peripheral arterial disease (PAD) and monitoring its response to therapy by measuring changes in microvessel alterations and perfusion variations.

DETAILED DESCRIPTION:
The clinical manifestations of peripheral arterial disease (PAD), regardless of etiology, are due to a lack of blood flow to the musculature relative to its metabolism, which results in pain in the affected muscle groups. PAD affecting the lower extremities causes claudication, cramping pain in the calf muscle, thigh or hip muscle induced by exercise. The initial test for evaluation of patients with claudication is ankle brachial index (ABI).

Therefore, a non-invasive and affordable US technique that can quantify blood perfusion and microvasculature density, without using contrast agent, will improve PAD detection in early stage and can monitor the disease progress as well as the treatment response. The investigators anticipate that our new cost-effective and non-invasive ultrasound perfusion technique offers a quantitative imaging of perfusion that would help separating PAD from non-PAD and monitor the disease progression and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers > 18 years old.
* Male and female volunteers with symptom of claudication and suspected peripheral arterial disease (PAD) who are scheduled for vascular testing.

Exclusion Criteria:

* Patients with gangrene.
* Patients with lower leg amputation.
* Having ulcer and any health condition that does not allow proper use of ultrasound scanning.
* People considered in "vulnerable" populations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Subject population will include n=300 symptomatic patients with claudication, at risk for PAD (150 abnormal ABI and 100 with normal ABI), male and female, age ≥18 years and are referred Mayo Clinic Vascular Center due to claudication or atypical leg symptoms for ABI examination. In addition to comparing to the group of Normal (symptomatic patients with normal resting and exercise ABI), the study will also include 50 healthy volunteers with normal ABI and with no history of smoking cardiovascular and metabolic disorders, including diabetes mellitus.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Aim 1: Determine the efficacy of ultrasonic perfusion imaging for early detection of PAD. The goal is to quantify the perfusion of cuff muscle in patients with lower leg claudication and compare the results to those obtained in healthy individuals | 4 yeas
  Perfusion density of the cuff muscle will be quantified by the new automatic ultrasound microvessel quantification technique and the resulting measurements will measure the outcome of this part of the study.

SECONDARY OUTCOMES:
Aim 2: Determine the efficacy of ultrasonic perfusion imaging for assessment of treatment response in PAD patients. The goal is to quantify the perfusion of the cuff muscle in PAD patients in 3 time points, 6 months, and every year after treatment. | 5 years
  At each time point after the treatment, the perfusion density of the cuff muscle will be quantified by the new automatic ultrasound microvessel quantification technique and the resulting measurements will measure the outcome of this part of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Azra Alizad, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT04755335/ICF_000.pdf